CLINICAL TRIAL: NCT03571516
Title: A Randomized, Open-label, 24-Week Safety, Efficacy, and Pharmacokinetic Study of Teduglutide in Infants 4 to 12 Months of Age With Short Bowel Syndrome Who Are Dependent on Parenteral Support
Brief Title: Safety, Efficacy and Pharmacokinetic Study of Teduglutide in Infants 4 to 12 Months of Age With Short Bowel Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHP633-301; 2017-003606-40 (EudraCT Number)
Record Dates: First submitted 2018-05-03; First posted 2018-06-27 (Actual); Results first posted 2021-04-08 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-04

CONDITIONS: Short Bowel Syndrome
Keywords: Short bowel syndrome; Teduglutide
MeSH Terms: conditions — Short Bowel Syndrome | interventions — teduglutide; Syringes; Needles

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Teduglutide (Experimental): Participants will receive 0.05 milligram per kilogram (mg/kg) subcutaneous (SC) injection of teduglutide into abdomen or into either the thigh or arm once daily (QD) in addition to standard medical therapy for 24 weeks.
  Interventions: Drug: Teduglutide; Other: Standard Medical Therapy; Device: Syringe; Device: Needle
- Standard of Care (SOC) (Other): Participants will receive standard medical therapy for 24 weeks.
  Interventions: Other: Standard Medical Therapy; Device: Syringe; Device: Needle

INTERVENTIONS:
Drug: Teduglutide — SC injection of 0.05 mg/kg teduglutide will be administered QD into abdomen or into either the thigh or arm for 24 weeks.
  Arms: Teduglutide
Other: Standard Medical Therapy — Standard medical therapy will be administered for 24 weeks.
Device: Syringe — Teduglutide will be administered using syringe (510k number: K980987).
Device: Needle — Teduglutide will be administered using needle (510k number: K021475).

SUMMARY:
The purpose of the study is to evaluate the safety, efficacy/pharmacodynamics (PD) and pharmacokinetics (PK) of teduglutide treatment in infants with short bowel syndrome (SBS) dependent on parenteral (PN) support.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent by the parent or legal guardian.
* Male or female infant 4 to 12 months corrected gestational age at screening.
* Weight at least 5 kilogram (kg) and weight-for-length Z-score greater than -2 at screening and baseline.
* Short bowel syndrome with dependence on parenteral support to provide at least 50% of fluid or caloric needs.
* Stable PN requirements for at least 1 month prior to screening, defined as a less than or equal to (<=) 10% change in the weight-normalized PN total fluid and caloric intake, despite attempts to wean PN, not withstanding transient instability for events such as sepsis or interruption of central venous access.
* Parent or legal guardian understands and is willing and able to fully adhere to study requirements as defined in this protocol.

Exclusion Criteria:

* Previous treatment with teduglutide.
* Intestinal malabsorption due to a genetic condition, such as cystic fibrosis, microvillus inclusion disease, etc.
* Severe, known dysmotility syndrome, such as pseudo-obstruction or persistent, severe, active gastroschisis-related dysmotility, that is the primary contributing factor to feeding intolerance and inability to reduce PN support, prior to screening. Dysmotility is defined as severe if it is expected to limit the advancement of enteral feeding.
* Inability to advance oral or enteral feeding due to lack of access to the gut, such as oral aversion in the absence of a feeding tube.
* Intestinal obstruction or clinically significant intestinal stenosis.
* Major gastrointestinal surgical intervention, such as serial transverse enteroplasty or major intestinal resection or anastomosis, within 3 months prior to screening or planned during the study period.
* Unstable cardiac disease.
* Renal dysfunction, defined as estimated glomerular filtration rate less than (<) 50 milliliter per minute (mL/min) per 1.73 square meter (m^2).
* Biliary obstruction, stenosis, or malformation.
* Clinically significant pancreatic disease.
* Severe hepatic dysfunction or portal hypertension, defined by at least 2 of the following parameters:

  1. International normalized ratio (INR) greater than (>) 1.5 not corrected with PN vitamin K
  2. Platelet count <100×10^3/ microliter (mcL) due to portal hypertension
  3. Presence of clinically significant gastric or esophageal varices
  4. Documented cirrhosis
* Persistent cholestasis defined as conjugated bilirubin >4 milligram per deciliter (mg/dL) (>68 micromoles per liter [mcmol/L]) over a 2 week period.
* More than 3 serious complications of intestinal failure (example [e.g.], catheter-associated bloodstream infections, interruption of nutrition due to feeding intolerance, catheter-associated thrombosis, severe fluid or electrolyte disturbances) within 1 month prior to or during screening.
* A history of cancer or a known cancer predisposition syndrome, such as juvenile polyposis or Beckwith-Wiedemann syndrome, or first degree relative with early onset of gastrointestinal cancer (including hepatobiliary and pancreatic cancers).
* Concurrent treatment with glucagon-like peptide-1 (GLP-1); glucagon-like peptide-2 (GLP-2); insulin-like growth factor-1 (IGF-1); growth hormone, somatostatin, or analogs of these hormones; or glutamine.
* Participation in a clinical study using an experimental drug within 3 months or 5.5 half-lives of the experimental drug, whichever is longer.
* Known or suspected intolerance or hypersensitivity to the investigational product, closely-related compounds, or any of the stated ingredients.
* Any condition, disease, illness, or circumstance that, in the investigator's opinion, puts the participant at any undue risk, prevents completion of the study, or interferes with analysis of the study results.

Ages: 4 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2018-08-31 (Actual); Primary Completion 2020-09-24 (Actual); Study Completion 2020-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Shire
Locations (8):
- Helsingin yliopistollinen keskussairaala, Helsinki, Finland
- France (2):
  - Groupe Hospitalier Pellegrin - Hôpital des Enfants, Bordeaux, Gironde
  - Hopital Jeanne de Flandre - CHRU Lille, Lille, Nord
- Ospedale Pediatrico Bambino Gesù, Roma, Italy
- United Kingdom (4):
  - Great Ormond Street Hospital for Children, London, Greater London
  - Royal Manchester Children's Hospital, Manchester, Greater Manchester
  - Alder Hey Childrens Hospital, Liverpool, Merseyside
  - Birmingham Children's Hospital, Birmingham, West Midlands

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data from this particular study will not be shared as there is a reasonable likelihood that individual patients could be re-identified (due to the limited number of study participants/study sites, …).

REFERENCES:
- [Derived] Chiba M, Masumoto K, Kaji T, Matsuura T, Morii M, Fagbemi A, Hill S, Pakarinen MP, Protheroe S, Urs A, Chen ST, Sakui S, Udagawa E, Wada M. Efficacy and Safety of Teduglutide in Infants and Children With Short Bowel Syndrome Dependent on Parenteral Support. J Pediatr Gastroenterol Nutr. 2023 Sep 1;77(3):339-346. doi: 10.1097/MPG.0000000000003867. Epub 2023 Jun 26. PMID 37364133
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b5fd94db2bf003ab4709b

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at Finland and United Kingdom between 31 August 2018 (first participant first visit) and 24 September 2020 (last participant last visit).
Pre-assignment Details: A total of 10 participants were enrolled into the study, of which 8 participants completed the study.
Groups:
- Teduglutide (TED): Participants (infants) 4 to 12 months of corrected gestational aged received 0.05 milligram per kilogram (mg/kg) of teduglutide subcutaneous (SC) injection QD in addition to standard medical therapy for 24 weeks.
- Standard of Care (SOC): Participants (infants) 4 to 12 months of corrected gestational aged received standard medical therapy for 24 weeks.
Period: Overall Study
Arm/Group | Teduglutide (TED) | Standard of Care (SOC)
Started | 5 | 5
Completed | 4 | 4
Not Completed | 1 | 1
Not completed — Severe diarrhea | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety set consisted of all participants who met the following criteria: Teduglutide treatment arm: participants who received at least 1 dose of teduglutide and had undergone at least 1 post baseline safety assessment; Standard of care treatment arm: participants who had undergone at least 1 post baseline safety assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Teduglutide (TED) | Standard of Care (SOC) | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: Months] | 8.5 (3.09) | 8.3 (2.65) | 8.4 (2.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 4 | 3 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 5 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 4 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieved At Least 20 Percent (%) Reduction From Baseline in Weight-normalized Parenteral Support (PS) Volume at End of Treatment/Early Termination (EOT/ET)
Description: Number of participants who achieved at least 20% reduction from baseline in weight-normalized PS volume at EOT/ET (up to Week 24) were reported. EOT/ET was defined as the last available visit after the date of first dose (or randomization in standard of care treatment group) during the 24-week treatment period.
Time Frame: Baseline, EOT/ET (up to Week 24)
Population: Intent-to-Treat (ITT) set consisted of all participants randomized in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Teduglutide (TED) | Standard of Care (SOC)
Number analyzed (Participants) | 5 | 5
Participants
  Diary Data: EOT/ET | 3 | 1
  Prescribed Data: EOT/ET | 3 | 3

2. Secondary Outcome: Plasma Concentration of Teduglutide at Nominal Time Points (Baseline at Pre-dose, and 1 Hour and 4 Hours Post-dose; 2 Hours Post-dose at Week 7)
Description: Mean plasma concentration of teduglutide was reported.
Time Frame: Baseline: Pre-dose,1, 4 hours post-dose, and 2 hours post-dose at Week 7
Population: Pharmacokinetic (PK) set consisted of all participants who received at least 1 dose of teduglutide and had at least 1 evaluable and interpretable post-dose PK concentration value. Here, the number of participants analyzed signifies participants who were evaluable for this outcome measure and number analyzed signifies participants who were evaluable at specific time point. Data was not planned to be collected and analyzed for SOC arm.
Measure: Median (Full Range); unit: Nanogram per milliliter (ng/mL)
Arm/Group | Teduglutide (TED)
Number analyzed (Participants) | 4
Nanogram per milliliter (ng/mL)
  Baseline: At Pre-dose | 0.00 [0.00 to 0.00]
  Baseline: At 1 hour: number analyzed (Participants) | 3
  Baseline: At 1 hour | 16.300 [7.25 to 25.70]
  Baseline: At 4 hours | 8.385 [3.86 to 22.5]
  Week 7: At 2 hours: number analyzed (Participants) | 2
  Week 7: At 2 hours | 16.950 [14.80 to 19.10]

3. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. TEAEs are defined as AEs that start or deteriorate on or after the date of the first dose of investigational product.
Time Frame: From start of study treatment up to end of study (EOS) (up to Week 28)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Teduglutide (TED) | Standard of Care (SOC)
Number analyzed (Participants) | 5 | 5
Participants | 5 | 5

4. Secondary Outcome: Change From Baseline in Body Weight Z-score at Week 24
Description: Body weight was measured using Z-score. Z-score was calculated as (observed value - median value of the reference population)/standard deviation value of reference population. A negative Z-score indicates values lower than the mean while a positive Z-score indicates values higher than the mean. Change from baseline in body weight Z-score at Week 24 was reported.
Time Frame: Baseline, Week 24
Population: Safety set consisted of all participants who met the following criteria: Teduglutide treatment arm: participants who received at least 1 dose of teduglutide and had undergone at least 1 post baseline safety assessment; Standard of care treatment arm: participants who had undergone at least 1 post baseline safety assessment. Here, the number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Teduglutide (TED) | Standard of Care (SOC)
Number analyzed (Participants) | 4 | 3
Z-score | -0.408 (0.377) | -0.289 (0.278)

5. Secondary Outcome: Change From Baseline in Length Z-Score at Week 24
Description: Length was measured using Z-score. Z-score was calculated as (observed value - median value of the reference population)/standard deviation value of reference population. A negative Z-score indicates values lower than the mean while a positive Z-score indicates values higher than the mean. Change from baseline in length Z-score at Week 24 was reported.
Time Frame: Baseline, Week 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Z-Score
Arm/Group | Teduglutide (TED) | Standard of Care (SOC)
Number analyzed (Participants) | 4 | 2
Z-Score | -0.274 (1.258) | -0.422 (0.384)

6. Secondary Outcome: Change From Baseline in Head Circumference Z-Score at Week 24
Description: Head circumference was measured using Z-score. Z-score was calculated as (observed value - median value of the reference population)/standard deviation value of reference population. A negative Z-score indicates values lower than the mean while a positive Z-score indicates values higher than the mean. Change from baseline in head circumference Z-score at Week 24 was reported.
Time Frame: Baseline, Week 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Z-Score
Arm/Group | Teduglutide (TED) | Standard of Care (SOC)
Number analyzed (Participants) | 4 | 2
Z-Score | -0.544 (0.446) | -0.167 (0.690)

7. Secondary Outcome: Change From Baseline in Weight-for-Length Z-Score at Week 24
Description: Weight-for-length was measured using Z-score. Z-score was calculated as (observed value - median value of the reference population)/standard deviation value of reference population. A negative Z-score indicates values lower than the mean while a positive Z-score indicates values higher than the mean. Change from baseline in weight-for-length Z-score at Week 24 was reported.
Time Frame: Baseline, Week 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Z-Score
Arm/Group | Teduglutide (TED) | Standard of Care (SOC)
Number analyzed (Participants) | 4 | 3
Z-Score | -0.447 (1.042) | -0.058 (0.992)

8. Secondary Outcome: Change From Baseline in Average Total Urine Output at Week 24
Description: Average total urine output was recorded over a 48-hour period of nutritional stability at Week 24 was reported. Here, milliliter per kilogram per day is abbreviated as mL/kg/day.
Time Frame: Baseline, Week 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mL/kg/day
Arm/Group | Teduglutide (TED) | Standard of Care (SOC)
Number analyzed (Participants) | 3 | 3
mL/kg/day | -0.61 (14.548) | 10.25 (17.383)

9. Secondary Outcome: Change From Baseline in Fecal Output at Week 24
Description: Change from baseline in the fecal output (average number of stools per day) at Week 24 was reported.
Time Frame: Baseline, Week 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Average number of stools per day
Arm/Group | Teduglutide (TED) | Standard of Care (SOC)
Number analyzed (Participants) | 3 | 3
Average number of stools per day | -3.33 (3.547) | 1.67 (1.756)

10. Secondary Outcome: Number of Participants With Positive Specific Antibodies to Teduglutide
Description: Number of participants with positive specific antibodies to teduglutide were used to summarize the presence of antibodies.
Time Frame: Baseline, EOS (up to week 28)
Population: Safety set: all participants who met the following criteria: Teduglutide treatment arm: participants who received at least 1 dose of teduglutide and undergone at least 1 post baseline safety assessment; Standard of care treatment arm: participants who had undergone at least 1 post baseline safety assessment. Here, number of participants analyzed signifies participants who were evaluable for this outcome measure. Data for this outcome was not planned to be collected and analyzed for SOC group.
Measure: Count of Participants; unit: Participants
Arm/Group | Teduglutide (TED)
Number analyzed (Participants) | 3
Participants | 0

11. Secondary Outcome: Number of Participants Who Achieved At Least 20 Percent (%) Reduction From Baseline in Weight-normalized Parenteral Support (PS) Caloric Intake at End of Treatment/Early Termination (EOT/ET)
Description: Number of participants who achieved at least 20% reduction from baseline in weight-normalized PS caloric intake at EOT/ET (up to Week 24) were reported. EOT/ET was defined as the last available visit after the date of first dose (or randomization in standard of care treatment group) during the 24-week treatment period.
Time Frame: Baseline, EOT/ET (up to Week 24)
Population: ITT set consisted of all participants randomized in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Teduglutide (TED) | Standard of Care (SOC)
Number analyzed (Participants) | 5 | 5
Participants
  Diary Data: EOT/ET | 3 | 1
  Prescribed Data: EOT/ET | 3 | 3

12. Secondary Outcome: Number of Participants Who Achieved 100 Percent (%) Reduction in Complete Weaning Off (Enteral Autonomy) Parenteral Support (PS) Volume at Week 24
Description: Number of participants who achieved 100% reduction in complete weaning off (enteral autonomy) PS volume at Week 24 were reported.
Time Frame: Week 24
Population: ITT set consisted of all participants randomized in the study. Here, the number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Teduglutide (TED) | Standard of Care (SOC)
Number analyzed (Participants) | 4 | 4
Participants | 0 | 0

13. Secondary Outcome: Number of Participants Who Achieved 100 Percent (%) Reduction in Complete Weaning Off (Enteral Autonomy) Parenteral Support (PS) Volume at End of Study (EOS)
Description: Number of participants who achieved 100% reduction in complete weaning off (enteral autonomy) PS volume at EOS (up to Week 28) were reported.
Time Frame: EOS (up to Week 28)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Teduglutide (TED) | Standard of Care (SOC)
Number analyzed (Participants) | 4 | 5
Participants | 0 | 0

14. Secondary Outcome: Change From Baseline in Weight-normalized Parenteral Support (PS) Volume at End of Treatment/Early Termination (EOT/ET)
Description: Change from baseline in weight-normalized PS volume at EOT/ET (up to Week 24) was reported. EOT/ET was defined as the last available visit after the date of first dose (or randomization in standard of care treatment group) during the 24-week treatment period.
Time Frame: Baseline, EOT/ET (up to Week 24)
Population: ITT set consisted of all participants randomized in the study. Here, the number analyzed signifies participants who were evaluable for this outcome at specific time points.
Measure: Mean (Standard Deviation); unit: mL/kg/day
Arm/Group | Teduglutide (TED) | Standard of Care (SOC)
Number analyzed (Participants) | 5 | 5
mL/kg/day
  Diary Data: EOT/ET: number analyzed (Participants) | 5 | 3
  Diary Data: EOT/ET | -21.54 (28.909) | -9.51 (7.497)
  Prescribed Data: EOT/ET | -22.90 (26.940) | -14.90 (12.323)

15. Secondary Outcome: Percent Change From Baseline in Weight-normalized Parenteral Support (PS) Volume at End of Treatment/Early Termination (EOT/ET)
Description: Percent change from baseline in weight-normalized PS volume at EOT/ET (up to Week 24) was reported. EOT/ET was defined as the last available visit after the date of first dose (or randomization in standard of care treatment group) during the 24-week treatment period.
Time Frame: Baseline, EOT/ET (up to Week 24)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Teduglutide (TED) | Standard of Care (SOC)
Number analyzed (Participants) | 5 | 5
Percent change
  Diary Data: EOT/ET: number analyzed (Participants) | 5 | 3
  Diary Data: EOT/ET | -24.77 (34.723) | -16.75 (16.392)
  Prescribed Data: EOT/ET | -27.28 (33.518) | -22.39 (17.198)

16. Secondary Outcome: Change From Baseline in Weight-normalized Parenteral Support (PS) Caloric Intake at End of Treatment/Early Termination (EOT/ET)
Description: Change from baseline in weight-normalized PS caloric intake at EOT/ET (up to Week 24) were reported. EOT/ET was defined as the last available visit after the date of first dose (or randomization in standard of care treatment group) during the 24-week treatment period. Here, kilo-calories per kilogram per day was abbreviated as (kcal/kg/day).
Time Frame: Baseline, EOT/ET (up to Week 24)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: kcal/kg/day
Arm/Group | Teduglutide (TED) | Standard of Care (SOC)
Number analyzed (Participants) | 5 | 5
kcal/kg/day
  Diary Data: EOT/ET: number analyzed (Participants) | 5 | 3
  Diary Data: EOT/ET | -16.14 (17.547) | -6.10 (10.386)
  Prescribed Data: EOT/ET | -15.31 (17.839) | -20.40 (21.024)

17. Secondary Outcome: Percent Change From Baseline in Weight-normalized Parenteral Support (PS) Caloric Intake at End of Treatment/Early Termination (EOT/ET)
Description: Percent change from baseline in weight-normalized PS caloric intake at EOT/ET (up to Week 24) were reported. EOT/ET was defined as the last available visit after the date of first dose (or randomization in standard of care treatment group) during the 24-week treatment period.
Time Frame: Baseline, EOT/ET (up to Week 24)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Teduglutide (TED) | Standard of Care (SOC)
Number analyzed (Participants) | 5 | 5
Percent change
  Diary Data: EOT/ET: number analyzed (Participants) | 5 | 3
  Diary Data: EOT/ET | -27.00 (29.473) | -13.68 (21.873)
  Prescribed Data: EOT/ET | -27.81 (30.777) | -38.86 (39.893)

18. Secondary Outcome: Change From Baseline in Weight-normalized Enteral Nutrition (EN) Volume at End of Treatment/Early Termination (EOT/ET)
Description: Change from baseline in weight-normalized EN volume at EOT/ET (up to Week 24) was reported. EOT/ET was defined as the last available visit after the date of first dose (or randomization in standard of care treatment group) during the 24-week treatment period.
Time Frame: Baseline, EOT/ET (up to Week 24)
Population: ITT set consisted of all participants randomized in the study. Here, the number of participants analyzed signifies participants who were evaluable for this outcome measure and number analyzed signifies participants who were evaluable at specific time point.
Measure: Mean (Standard Deviation); unit: mL/kg/day
Arm/Group | Teduglutide (TED) | Standard of Care (SOC)
Number analyzed (Participants) | 4 | 5
mL/kg/day
  Diary Data: EOT/ET: number analyzed (Participants) | 4 | 3
  Diary Data: EOT/ET | 16.14 (18.683) | -15.25 (31.496)
  Prescribed Data: EOT/ET | -1.28 (2.563) | 2.27 (22.232)

19. Secondary Outcome: Percent Change From Baseline in Weight-normalized Enteral Nutrition (EN) Volume at End of Treatment/Early Termination (EOT/ET)
Description: Percent change from baseline in weight-normalized EN volume at EOT/ET (up to Week 24) was reported. EOT/ET was defined as the last available visit after the date of first dose (or randomization in standard of care treatment group) during the 24-week treatment period.
Time Frame: Baseline, EOT/ET (up to Week 24)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Teduglutide (TED) | Standard of Care (SOC)
Number analyzed (Participants) | 2 | 4
Percent change
  Diary Data: EOT/ET: number analyzed (Participants) | 2 | 2
  Diary Data: EOT/ET | 273.20 (246.784) | -44.25 (78.847)
  Prescribed Data: EOT/ET: number analyzed (Participants) | 1 | 4
  Prescribed Data: EOT/ET | -16.40 (NA) — Here, standard deviation was not analyzed due to single participant. | 14.80 (69.834)

20. Secondary Outcome: Change From Baseline in Weight-normalized Enteral Nutrition (EN) Caloric Intake at End of Treatment/Early Termination (EOT/ET)
Description: Change from baseline in weight-normalized EN caloric intake at EOT/ET (up to Week 24) were reported. EOT/ET was defined as the last available visit after the date of first dose (or randomization in standard of care treatment group) during the 24-week treatment period.
Time Frame: Baseline, EOT/ET (up to Week 24)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: kcal/kg/day
Arm/Group | Teduglutide (TED) | Standard of Care (SOC)
Number analyzed (Participants) | 4 | 5
kcal/kg/day
  Diary Data: EOT/ET: number analyzed (Participants) | 4 | 3
  Diary Data: EOT/ET | 9.08 (10.662) | -9.38 (21.402)
  Prescribed Data: EOT/ET | -1.15 (2.306) | 3.11 (16.285)

21. Secondary Outcome: Percent Change From Baseline in Weight-normalized Enteral Nutrition (EN) Caloric Intake at End of Treatment/Early Termination (EOT/ET)
Description: Percent change from baseline in weight-normalized EN caloric intake at EOT/ET (up to Week 24) were reported. EOT/ET was defined as the last available visit after the date of first dose (or randomization in standard of care treatment group) during the 24-week treatment period.
Time Frame: Baseline, EOT/ET (up to Week 24)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Teduglutide (TED) | Standard of Care (SOC)
Number analyzed (Participants) | 2 | 4
Percent change
  Diary Data: EOT/ET: number analyzed (Participants) | 2 | 2
  Diary Data: EOT/ET | 207.06 (153.159) | -44.25 (78.847)
  Prescribed Data: EOT/ET: number analyzed (Participants) | 1 | 4
  Prescribed Data: EOT/ET | -16.40 (NA) — Here, standard deviation was not analyzed due to single participant. | 24.18 (78.115)

22. Secondary Outcome: Number of Participants Who Achieved At Least 20 Percent (%) Increase From Baseline in Weight-normalized Enteral Nutrition (EN) Volume at End of Treatment/Early Termination (EOT/ET)
Description: Number of participants who achieved at least 20% increase from baseline in weight-normalized EN volume at EOT/ET was reported. EOT/ET was defined as the last available visit after the date of first dose (or randomization in standard of care treatment group) during the 24-week treatment period.
Time Frame: Baseline, EOT/ET (up to Week 24)
Population: ITT set consisted of all participants randomized in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Teduglutide (TED) | Standard of Care (SOC)
Number analyzed (Participants) | 5 | 5
Participants
  Diary Data: EOT/ET | 2 | 0
  Prescribed Data: EOT/ET | 0 | 2

23. Secondary Outcome: Number of Participants Who Achieved At Least 20 Percent (%) Increase From Baseline in Weight-normalized Enteral Nutrition (EN) Caloric Intake at End of Treatment/Early Termination (EOT/ET)
Description: Number of participants who achieved at least 20% increase from baseline in weight-normalized EN caloric intake at EOT/ET was reported. EOT/ET was defined as the last available visit after the date of first dose (or randomization in standard of care treatment group) during the 24-week treatment period.
Time Frame: Baseline, EOT/ET (up to Week 24)
Population: ITT set consisted of all participants randomized in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Teduglutide (TED) | Standard of Care (SOC)
Number analyzed (Participants) | 5 | 5
Participants
  Diary Data: EOT/ET | 2 | 0
  Prescribed Data: EOT/ET | 0 | 2

ADVERSE EVENTS:
Time Frame: From start of study treatment up to end of study (EOS) (up to Week 28)
Arm/Group | Teduglutide (TED) | Standard of Care (SOC)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 4/5 | 3/5
Other Adverse Events (participants affected / at risk) | 5/5 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Teduglutide (TED) (N=5) | Standard of Care (SOC) (N=5)
Pyrexia (General disorders) | 1 (2) | 0 (0)
Immunisation reaction (Immune system disorders) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 2 (2)
Transaminases increased (Investigations) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1)
Device breakage (Product Issues) | 1 (1) | 0 (0)
Device leakage (Product Issues) | 1 (1) | 0 (0)
Device occlusion (Product Issues) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Teduglutide (TED) (N=5) | Standard of Care (SOC) (N=5)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (3) | 0 (0)
Abnormal faeces (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucous stools (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retching (Gastrointestinal disorders) | 1 (1) | 0 (0)
Teething (Gastrointestinal disorders) | 0 (0) | 2 (3)
Vomiting (Gastrointestinal disorders) | 3 (8) | 1 (2)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Secretion discharge (General disorders) | 1 (1) | 0 (0)
Gastroenteritis norovirus (Infections and infestations) | 1 (1) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 0 (0) | 1 (1)
Medical device site infection (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2)
Viral infection (Infections and infestations) | 1 (1) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lip injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (2) | 0 (0)
Blood iron decreased (Investigations) | 0 (0) | 1 (1)
Faecal volume increased (Investigations) | 1 (1) | 0 (0)
Respiratory rate increased (Investigations) | 0 (0) | 1 (1)
Serum ferritin decreased (Investigations) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 1 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypophagia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Device breakage (Product Issues) | 1 (1) | 1 (1)
Device occlusion (Product Issues) | 1 (1) | 0 (0)
Irritability (Psychiatric disorders) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (2):
  • Study Protocol (2019-12-17): https://cdn.clinicaltrials.gov/large-docs/16/NCT03571516/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-24): https://cdn.clinicaltrials.gov/large-docs/16/NCT03571516/SAP_001.pdf